CLINICAL TRIAL: NCT07002996
Title: Spatial Memory Training and Cognitive Function
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Douglas Mental Health University Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Véronique Bohbot, Professor, Douglas Mental Health University Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Auto-SMIP-001; 488505 (Other Grant/Funding Number: Canadian Institutes for Health Research)
Record Dates: First submitted 2025-05-07; First posted 2025-06-04 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Mild Cognitive Impairment
Keywords: Memory; Spatial Memory; Hippocampus; Cognitive Training; Cognitive Decline; Aging
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Co-investigators
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SMIP (Experimental): Spatial Memory Intervention Program
  Interventions: Behavioral: SMIP
- Control (Placebo Comparator): The control group will receive no intervention between baseline and follow-up.
  Interventions: Other: No intervention

INTERVENTIONS:
Behavioral: SMIP — Participants will undergo a 3-month-long regimen of 60 minutes spatial memory training sessions held twice a week, consisting of a series of computerized virtual reality tasks.
  Arms: SMIP
Other: No intervention — Control participants will not receive spatial memory intervention training. They will watch documentaries and then complete multiple choice quizzes on its content to ensure they are paying attention. The placebo condition will match the experimental condition in terms of duration and visit frequency.
  Arms: Control

SUMMARY:
Mild cognitive impairment (MCI) is often considered a transitional stage between normal aging and dementia, particularly Alzheimer's disease (AD). Patients with MCI have subjective memory complaints corroborated by standard neuropsychological tests but remain functionally autonomous. One of the first brain regions to show AD pathology is the hippocampus (HPC). Reduction in HPC volume is a strong predictor of AD dementia. Therefore, improvement or restoration of HPC structure and function is thus an attractive target for improvement in memory and AD prevention strategies. In the current study, the investigators propose to examine the effects of a 3-month long spatial memory program on spatial memory and the hippocampus in patients diagnosed with MCI. Neuropsychological tests are also administered before and after the training to assess the effects of the intervention on cognition. In our previous research, the investigators have shown that spatial memory intervention program (SMIP) improves cognition and hippocampal based spatial memory compared to controls.

DETAILED DESCRIPTION:
The hippocampus (HPC) is a labile structure capable of neurogenesis and synaptic plasticity throughout the lifespan, which is thought to underlie its role in learning and memory, particularly of autobiographical and spatial events. Numerous studies have associated the integrity of the hippocampus with performance in way-finding. In fact, it has been demonstrated that individuals who acquired a cognitive representation of an environment with greater ease possessed more hippocampal gray matter, which was positively correlated with experience. These and other similar studies have suggested that the hippocampus' ability to process spatial memory can be modulated by experience or practice.

Studies have demonstrated increased grey matter in the HPC of both young and older human adults as a function of memory training. Interestingly, the HPC shows signs of neurogenesis across the entire lifespan and, in adult primates, this HPC neurogenesis can be stimulated through learning and memory programs that increase HPC cellular survival. Similar training programs may thus enhance HPC cellular survival in Mild Cognitive Impairment (MCI) patients by focusing on the region where the pathology first emerges. While several memory intervention studies have shown success in alleviating memory impairments in participants with subjective cognitive impairment, MCI, and in patients with Alzheimer's disease by presumably affecting the HPC, this has not yet been supported by brain imaging or assessment. By contrast, using virtual reality-based tools, the investigators have developed an innovative learning and memory program. In previous research with healthy older adults, the investigators have shown that spatial memory intervention program (SMIP) improves cognition and hippocampal-based spatial memory compared to controls. In addition, the investigators have shown a positive impact of such training on HPC grey matter. These grey matter changes in the HPC were beneficial to healthy cognition as they correlated to improvements in memory.

In the current study, the investigators propose a randomized controlled trial comparing the effects of a 12-week spatial memory intervention to an active control condition. The design will be stratified according to age, education, and sex. After an eligibility assessment at baseline, participants meeting inclusion criteria will be randomly allocated to one of the two groups with a 50% probability of being enrolled in either a spatial memory intervention or an active placebo condition. In addition, participants will be given a pre-training psychometric battery, which will be repeated twice during two post-training sessions (at one- and 26 weeks post-training) to assess cognition, daily functioning, stress, health, physical activity, quality of life, and self-esteem. The battery will also include independent computerized spatial memory tests assessing the generalization of cognitive improvement in the spatial domain, as well as paper and pencil memory tests described below.

ELIGIBILITY:
Inclusion Criteria:

1. Age 55 years and above.
2. Primary language is English or French.
3. Individuals having received a diagnosis of Mild Cognitive Impairment (MCI).

Exclusion Criteria:

1. Self-reported having either of the following:

   Current post-traumatic stress disorder and/or generalized anxiety disorder; Substance use disorder; Significant heart disease (i.e., stroke occurring during 5 years prior to study assessment or cardiac disease non-stabilized with medication); Severe Depression, or a Geriatric Depression Scale (GDS) score greater than 12; Current insomnia disorder.
2. Current medications for sleep problems, or use of medications that affect sleep.
3. Use of antidepressant and anti-anxiety medication for less than 3 months prior to study entry.
4. Use of analgesics with codeine (or other opioids).
5. Use of antipsychotic medication (past or current).
6. Having undergone brain surgery or ECT.
7. Self-reported colour-blindness.
8. General anesthesia in the past year.
9. Current smoker.
10. Suspected or confirmed traumatic brain injury during the last 24 months.
11. Motion sickness or intolerant to virtual reality tasks.
12. Cholesterol or hypertension medication for less than 3 months or changes expected within the next 9 months.
13. History or presence of neurological or psychiatric disorders (other than MCI) that in the opinion of the investigator may compromise patient safety or study objectives.
14. Current severe medical conditions (e.g. untreated diabetes, cancer) that in the opinion of the investigator may compromise patient safety or study objectives.
15. For female participants, severe menopausal symptoms, including hot flashes (determined from the Greene climacteric scale - any participants scoring over 15 is excluded).
16. Use of computer games that are designed to help with memory or general cognition.
17. Presence of any medical or psychological condition that, in the opinion of the principal investigator, may compromise the study objectives.
18. Presence of contra-indications for MRI scanning.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-06-15 (Actual); Primary Completion 2030-09-30 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in hippocampal atrophy score using SNIPE (Scoring by Non-local Image Patch Estimator) | From study entry to Week 16 in hippocampus SNIPE grading.
  Hippocampal atrophy will be assessed by applying the SNIPE algorithm to T1-weighted structural MRI scans. The SNIPE score quantifies similarity of hippocampal image patches to those found in Alzheimer's disease (AD) patients and cognitively healthy controls, providing a continuous score ranging from -1 (AD-like) to +1 (control-like). Change in SNIPE score from baseline to post-treatment will be used to evaluate the effect of the intervention on neurodegeneration.

SECONDARY OUTCOMES:
Hippocampal volume. | From study entry to weeks 16 and 41.
  Changes in hippocampal volume as determined by structural magnetic resonance imaging (MRI).
Change in hippocampal atrophy score using SNIPE (Scoring by Non-local Image Patch Estimator) at 41 weeks post-study entry. | From study entry to Week 41.
  Hippocampal atrophy will be assessed by applying the SNIPE algorithm to T1-weighted structural MRI scans. The SNIPE score quantifies similarity of hippocampal image patches to those found in Alzheimer's disease (AD) patients and cognitively healthy controls, providing a continuous score ranging from -1 (AD-like) to +1 (control-like). Change in SNIPE score from baseline to post-treatment will be used to evaluate the effect of the intervention on neurodegeneration.
Changes in spatial memory performance. | From study entry to weeks 15 and 40.
  Changes in spatial memory performance will be assessed according to the Functional Spatial Abilities Questionnaire (FSAQ), a 12-item self-report tool developed to assess spatial orientation and navigation abilities. Respondents rate their difficulty for a series of tasks. The total score, ranging from 12 to 36, is calculated by summing the individual item scores, with higher total scores indicating greater impairment in functional spatial abilities.
Changes in spatial memory performance: radial maze task. | From study entry to weeks 15 and 40.
  The 4-on-8 virtual maze is a computerized task which will be used to investigate spontaneous strategies used by participants. Participants have to find 4 hidden objects in an 8-arm radial-maze. Performance is measured in terms of errors committed.
Changes in spatial memory performance: Paired arms radial maze task. | From study entry to weeks 15 and 40.
  Changes in spatial memory performance will be assessed according to the Concurrent Spatial Discrimination Learning Task (CSDLT). Participants complete a virtual reality program in which they are required to find a target object among a pair of arms presented simultaneously in a 12-arm radial maze. Performance is measured in terms of errors committed.
Changes in spatial memory performance: Way-finding task. | From study entry to weeks 15 and 40.
  Participants are required to locate objects located in a virtual space. Performance is measured in terms of errors committed.
Changes in verbal learning performance | From study entry to weeks 15 and 40.
  Rey Auditory Verbal Learning Task: participants are required to learn a list of 15 words via multiple trials, with immediate recall, delayed recall and recognition components.
Change in visual memory performance. | From study entry to weeks 15 and 40.
  Visual memory performance is evaluated according immediate and delayed recall in the Rey and Taylors complex figures tests (alternate versions used across visits).
Changes in general cognition. | From study entry to weeks 15 and 40.
  General cognition is evaluated using the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS). The battery, a standardized neuropsychological assessment used to evaluate cognitive functioning in adults, yields scores ranging from 40 to 160, with higher scores reflecting greater functioning.
Changes in general intelligence level. | From study entry to weeks 15 and 40.
  Changes in general intelligence will be evaluated according to the Test of Nonverbal Intelligence, Third Edition (TONI-3), which is a standardized assessment designed to measure abstract reasoning and problem-solving abilities without relying on verbal communication or motor skills. The TONI-3 consists of 45 items, with a raw score range of 0 to 45, with higher scores reflecting greater intelligence.
Changes in selective attention performance. | From study entry to weeks 15 and 40.
  Selective attention performance will be assessed according to the Stroop Neuropsychological Screening Test (adult version).
Changes in visuomotor working memory performance: Trail making | From study entry to weeks 15 and 40.
  Changes in visual spatial motor performance will be assessed according to the Trail-making test of the D-KEF battery.
Changes in self-reported sense of direction: Santa Barbara Sense of Direction Scale | From study entry to weeks 15 and 40.
  Changes in self-reported sense of direction will be ascertained according to the Santa Barbara Sense of Direction Scale (SBSDS), a 15-item self-report tool developed to assess navigational and spatial abilities. Respondents rate agreement for a series of spatial navigation related statements . The total score, ranging from 1 to 7, is calculated by summing the individual item scores and averageing them, with higher total scores indicating greater sense of direction.
Changes in self-reported sense of direction: Sense of Direction Questionnaire- Short-Form | From study entry to weeks 15 and 40.
  Changes in self-reported sense of direction will be ascertained according to the Sense of Direction Questionnaire- Short-Form (SDQ-S), a 15-item self-report tool developed to assess awareness of orientation and memory for usual spatial behavior. Respondents rate agreement for a series of spatial navigation related statements. The total score, ranging from 17 to 75, is calculated by summing the individual item scores, with higher total scores indicating greater sense of direction.
Changes in self-reported well-being. | From study entry to weeks 15 and 40.
  Changes in self-reported well-being will be assessed according to the General Well Being Schedule, which includes positive and negative questions across six dimensions: well-being, self-control, vitality, depression, anxiety, and general health. Scores on this scale vary from 0 to 110, with higher scores representing better perceived well-being.
Changes in self-reported meta-memory. | From study entry to weeks 15 and 40.
  Changes in self-reported meta-memory will be evaluated according to the Multifactorial Memory Questionnaire Strategies (MMQ-Strategies), a 19-item tool developped to measures satisfaction with memory functioning, self-reported use of memory strategies, and self-appraisal of memory ability. The score, ranging from 0 to 76, is calculated by summing the individual item scores, with higher scores indicating greater use of memory strategies.
Changes in self-reported attention, memory, and cognition in everyday life. | From study entry to weeks 15 and 40.
  Changes in self-reported attention, memory, and cognition in everyday life will be measured according to the Cognitive Failures Questionnaire (CFQ), a 25-item self-report measure that assesses everyday cognitive failures or minor mistakes over the past 6 months. Respondents rate how often each mistake occurs. The score, ranging from 0 to 100, is calculated by summing the individual item scores, with higher scores indicating more cognitive failures.
Changes in self-reported quality of life. | From study entry to weeks 15 and 40.
  Changes in self-reported quality of life will be determined according to the 36-Item Short Form Health Survey (SF-36), a self-report survey designed to assess mental and physical health impact on quality of life. The scale is divided in 6 subscales, physical functioning, physical limitation, emotional well-being and emotional limitations, energy/fatigue, social functioning, pain and general health. Each subscales ranges from 0 to 100, with higher score reflecting better quality of life.
Changes in perceived stress. | From study entry to weeks 15 and 40.
  Changes in perceived stress will be evaluated according to the Perceived Stress Scale, a 14-item scale that assess how different situations affect feelings and perceived stress. Respondents rate how often feelings and thoughts occurred during the last month. The scale ranges from 0 to 56 is calculated by summing the individual item scores, with a higher score indicating higher perceived stress.
Changes in mindfulness. | From study entry to weeks 15 and 40.
  Changes in mindfulness will be assessed according to the Five-Facet Mindfulness Questionnaire, a 39-item tool developed to assess an individual's mindfulness and self-awareness. Respondents rate statements about mindfulness. The overall score ranging from 39 to 195, is calculated by summing the individual item scores, with higher scores reflecting more mindfulness.
Changes in State-Trait Anxiety. | From study entry to weeks 15 and 40.
  Changes in state-train anxiety will be ascertained according to the State-Trait Anxiety Inventory, a 40-item inventory developed to assess state and trait anxiety. Respondents rate state and trait statements about how they feel in the present moment and in general. The score, ranging from 40 to 160, is calculated by summing the individual item scores, with higher scores reflecting higher anxiety.
Changes in knowledge, usage, and opinions regarding GPS technology. | From study entry to weeks 15 and 40.
  Changes in users' knowledge, usage, and opinions regarding GPS technology will be assessed using the Global Positioning System (GPS) questionnaire, a tool developped to assess GPS dependence and frequency of use. The total score ranging from 23 to 115 is calculated by summing the individual item scores, with higher total scores indicating greater GPS use.
Changes in ability to perform activities in daily living. | From study entry to weeks 15 and 40.
  Changes in activities in daily living will be assessed according to an abbreviated version of the DAD scale (disability assessment for dementia: DAD-6), an instrument for detection of loss of autonomy. Respondents answer questions related to activities of daily living. The score, ranging from 0 to 18, is calculated by summing the individual item scores, with higher scores indicating higher autonomy.
Changes in cognitive reserve level. | From study entry to weeks 15 and 40.
  Changes in cognitive reserve level will be assessed according to the Cognitive Reserve Index Questionnaire, a questionnaire designed to measure an individual's capacity to compensate for susceptibility to cognitive impairment associated with age. The total score has a mean of 100 and a standard deviation of 15, with higher scores indicating more cognitive reserve.
Changes in physical activity level. | From study entry to weeks 15 and 40.
  Changes in physical activity level will be measured according to the Global Physical Activity Questionnaire, which was developed for assessing physical activity participation in three settings (Activity at work, Travel to and from places, and Recreational activities) as well as sedentary behavior. The score, ranging from 0 to 100, is calculated by averaging daily percentage of total physical activity, with higher scores indicating more physical activity.
Changes in Mini Mental State Exam score. | From study entry to weeks 15 and 40.
  Changes in cognition will be evaluated according to the Mini Mental State Exam scores, using 11 questions that assess five areas of cognitive function: orientation, registration, attention and calculation, recall, and language. The score, ranging from 0 to 30, is calculated by summing the individual item scores, with higher scores indicating less cognitive impairment.
Changes in Montreal Cognitive Assessment scale scores. | From study entry to weeks 15 and 40.
  Changes in cognition according to the Montreal Cognitive Assessment (MoCA) scale, a screening tool used to assess mild cognitive impairment. Respondents are evaluated on various cognitive domains, including attention, memory, language, and executive functions. The score, ranging from 0 to 30, is calculated by summing the sections scores, where a score of 26 or above is considered normal.
Changes in autobiographical memory. | From study entry to weeks 15 and 40.
  Changes in autobiographical memory will be assessed according to the Survey of Autobiographical Memory, a 26-item self-report tool developed to assess autobiographical memory capacities. Respondents rate statements about their autobiographical memory. The scale ranging from 26 to 130 is calculated by summing the individual item scores, with higher scores reflecting better autobiographical memory.
Changes in verbal fluency performance. | From study entry to weeks 15 and 40.
  Changes in verbal fluency performance will be assessed according to the D-KEFs verbal fluency test.
Changes in quality of life. | From study entry to weeks 15 and 40.
  Changes in quality of life level will be assessed according to the Quality of life scale (long version), a tool developed to assess quality of life. The scale, ranging from 0 to 100, is calculated by summing the individual item scores, with higher scores representing better quality of life.
Changes in self-reported memory ability. | From study entry to weeks 15 and 40.
  Changes in self-reported memory ability will be assessed according to the Self-Report Memory Scale (Memory Assessment Clinics Self-Rating Scale), a 42-item self-report scale that assesses the ability to remember. Respondents rate statement about their ability to remember. The scale, ranging from 42 to 210, is calculated by summing the individual item scores, with higher scores reflecting better ability to remember.
Changes in self-reported memory complaint. | From study entry to weeks 15 and 40.
  Changes in self-reported memory complaint will be assessed according to the Auto-administered memory questionnaire, a 64-item french scale developed to assess memory complaints. The scale, ranging from 64 to 384, is calculated by summing the individual item scores, with higher scores reflecting greater subjective memory complaints.
Changes in self-esteem. | From study entry to weeks 15 and 40.
  Changes in self-esteem will be measured according the Rosenberg Self-Esteem Questionnaire, a 10-item scale developed to assess self-esteem. The scale, ranging from 10 to 40, is calculated by summing the individual item scores, with higher scores reflecting higher self-esteem.
Changes in impulsivity. | From study entry to weeks 15 and 40.
  Changes in impulsivity will be measured according to the Barrat Impulsivity Scale, a 30-item scale developed to assess impulsivity. The scale, ranging from 30 to 120, is calculated by summing the individual item scores, with higher scores reflecting higher impulsivity.
Impact of spatial memory training on self-reported memory performance. | From study entry to weeks 15 and 40.
  Changes in self-reported memory scores for all questionnaires metionned above will be compared across groups.
Changes in inhibitory control. | From study entry to weeks 15 and 40.
  Changes in inhibitory control will be assessed according to the go-no-go test.
Effect of spatial memory training on subjective memory. | From study entry to weeks 15 and 40.
  Changes in daily life aspects will be assessed according to the Spatial Memory Training Program(SMTP) Subjective Interview Questionnaire, an in-house self-report questionnaire designed to measure subjective memory changes, mood changes as well as any other subjective changes that the participant experienced since the beginning of the training. The scale, ranging from 12 to 58, is calculated by summing the individual item scores, with higher scores representing more positive changes.

CONTACTS AND LOCATIONS:
Overall Officials: Véronique Bohbot, Ph.D., Principal Investigator — Douglas Mental Health University Institute
Locations (1):
- Douglas Mental Health University Institute, Verdun, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bohbot VD, Iaria G, Petrides M. Hippocampal function and spatial memory: evidence from functional neuroimaging in healthy participants and performance of patients with medial temporal lobe resections. Neuropsychology. 2004 Jul;18(3):418-25. doi: 10.1037/0894-4105.18.3.418. PMID 15291720
- [Background] Bohbot VD, Lerch J, Thorndycraft B, Iaria G, Zijdenbos AP. Gray matter differences correlate with spontaneous strategies in a human virtual navigation task. J Neurosci. 2007 Sep 19;27(38):10078-83. doi: 10.1523/JNEUROSCI.1763-07.2007. PMID 17881514
- [Background] Iaria G, Petrides M, Dagher A, Pike B, Bohbot VD. Cognitive strategies dependent on the hippocampus and caudate nucleus in human navigation: variability and change with practice. J Neurosci. 2003 Jul 2;23(13):5945-52. doi: 10.1523/JNEUROSCI.23-13-05945.2003. PMID 12843299